CLINICAL TRIAL: NCT04735991
Title: A Real-world Clinical Study Evaluating the Quality of Life in Family Members of Colorectal Cancer Patients Based on a Whole Course Chronic Disease Management System for Cancer Patients' Family
Brief Title: A Real-world Clinical Study of Kapok Initiative
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment process is affected by the coronavirus pandemic.
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: QTC care (Unknown)
Responsible Party: Principal Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LZMMH-2020
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The patient's family members need to fill in the family member quality of life questionnaire during the screening and follow-up period. They are able to contact the doctor for questions in terms of medical treatment.
- Study group (Experimental): The family members of the patients need to fill in the family member quality of life questionnaire during the screening period and follow-up period, and are involved in an interactive management program on the mobile terminal, full participation required.
  Interventions: Behavioral: Kapok Initiative

INTERVENTIONS:
Behavioral: Kapok Initiative — The detailed process is:
  1. After randomization, the Kapok assistant will contact the patient's family
  2. The family of the patient joins the "Kapok Initiative". They will participate in a 60-minute training program for 27 days, which is taught online by experts; The contents of the lectures are as follows: 1) Doctors are also mortal; 2) New medicines and new therapies; 3) Alternative therapies; 4) Don't panic during the operation; 5) Pain relief; 6) Side effects of treatment; 8) About the truth; 9) New topics; 10) Anti-cancer cost-effectiveness; 11) Medical insurance; 12) Commercial medical insurance; 13) Exercise and rehabilitation; 14) Nutrition and Foods to increase leukocytes level; 15) Long-term persistence; 16) Acceptance Change; 17) Two new roles; 18) Future expectation.
  Arms: Study group

SUMMARY:
This study is a prospective and effective research study. The aim is to assess the difference in the quality of life of the family members of patients with colorectal cancer after application of follow-up disease management using mobile network terminals and routine clinical treatment follow-up management. The hypothesis is that the application of mobile-based disease management system significantly improves the quality of life of the patients' family members, thereby improving the quality of life of the patients' families.

Approximately 100 families of colorectal cancer patients who had been diagnosed as high-risk stage II or stage III and required adjuvant chemotherapy XELOX regimen within 6 months after initial diagnosis were randomly assigned to the control and study groups at a 1: 1 ratio, with approximately 50 cases in the control group and about 50 patients in the study group. The reason for choosing these tumors is because the patients with these tumors will present a series of clinical symptoms during the treatment, which requires family members to take care of them. All patient and their family demographics, questionnaires on quality of life of patient's family, adverse events and other information will be collected.

The study uses a network-centric randomization system. In the randomization process, stratified randomization will be carried out according to the education level of the patient's family members (junior college degree or above vs. below college degree). The family members of the patients participating in the study will be randomly assigned to the tumor patient management platform or clinical routine treatment follow-up group.

Family members of all patients will be followed up to 2 months after randomization, or withdrew from the study (with the preceding events as the end point). Unless the patient's family member withdraws from the study, lost to follow-up, or the study is terminated, the patient is considered to be in the study. Family members of patients who are randomly assigned to the full management platform need to participate in a 60 minutes concentrated training session for 27 days, taught by experts online. The content of the lectures includes medical treatment guidelines, pain relief, family rehabilitation, family communication, family roles, early screening prevention, Medical insurance and other aspects. The contents of the online courses are: 1) Doctors are also mortal; 2) New medicines and new therapies; 3) Alternative therapies; 4) Don't panic during the operation; 5) Pain relief; 6) Side effects of treatment; 8) About the truth; 9) New topics; 10) Anti-cancer cost-effectiveness; 11) Medical insurance; 12) Commercial medical insurance; 13) Exercise and rehabilitation; 14) Nutrition and Foods to increase leukocytes level ; 15) Long-term persistence; 16) Acceptance Change; 17) Two new roles; 18) Future expectation.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subject: The main family members caring for patients are ≥18 and ≤65 years old;
* (2) Family members of patients who can understand the purpose of the study, voluntarily participate and sign an informed consent form, and are willing to complete follow-up as required by the protocol;
* (3) Family members of colorectal cancer patients who need to receive adjuvant chemotherapy XELOX regimen within 6 months after initial diagnosis of high-risk stage II or stage III

Exclusion Criteria:

* (1) Patient life expectancy is less than 3 months
* (2) Family members of patients cannot use electronic mobile products
* (3) The family of the patient has a history of malignant tumors or other serious diseases
* (4) Family members of patients are considered unsuitable by the researcher

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
To assess the difference in the quality of life of the family members of patients with colorectal cancer after application of follow-up disease management using mobile network terminals and routine clinical treatment follow-up management. | 1 Month
  First of all, The Cronbach's α coefficient of the QOLLTI-F family quality of life questionnaire that is used in this study will be calculated; then the minimum, maximum, median (quartile) and mean (standard deviation) of the quality of life scores of the family members of the study group and the control group will be determined; finally we will use t test to compare the scores to investigate whether there is a difference in the quality of life score between two groups; in order to eliminate the influence of confounding factors (such as age, gender, education level, etc.) on the main research results, several common influencing factors will be selected to construct a covariance analysis regression model to assess whether the intervention strategy of this study has an impact on the quality of life of patients' family members.

SECONDARY OUTCOMES:
To assess the difference in quality of life of subjects (family of patients) with different educational levels | 1 Month
  Patients' families are grouped based on their educational level, and the minimum, maximum, median (quartile), and mean (standard deviation) of the scores of quality of life questionnaire of each group will be calculated; Analysis of variance will be used to compare whether there are differences in the quality of life scores of patients' families among different education levels. If a general difference occurs, the Bonferroni method will be used to further perform multiple comparisons. At the same time, the Kruskal-Wallis rank-sum test will be used to compare the overall differences between the groups and the Steel-Dwass-Critchlow-Fligner test will be used for further multiple comparisons.
To assess the difference in the quality of life of the relationship between the subject (patient's family member) and the patient | 1 Month
  The subjects will be grouped according to the relationship between the subjects (families of patients) and patients. The minimum, maximum, median (quartile), and mean (standard deviation) of the scores of quality of life questionnaire of each group will be calculated; Analysis of variance will be used to compare whether there are differences in the quality of life scores of patients' families among different education levels. If a general difference occurs, the Bonferroni method will be used to further perform multiple comparisons. At the same time, the Kruskal-Wallis rank-sum test will be used to compare the overall differences between the groups and the Steel-Dwass-Critchlow-Fligner test will be used for further multiple comparisons.
To assess the difference in quality of life of the subjects (family of patients) with difference length of time spent taking care of the patients daily | 1 Month
  The minimum, maximum, median (quartile), and mean (standard deviation) of the scores of quality of life questionnaire based on difference length of time spent on daily care will be calculated; Analysis of variance will be used to compare whether there are differences in the quality of life scores of patients' families among different education levels. If a general difference occurs, the Bonferroni method will be used to further perform multiple comparisons. At the same time, the Kruskal-Wallis rank-sum test will be used to compare the overall differences between the groups and the Steel-Dwass-Critchlow-Fligner test will be used for further multiple comparisons.
To assess the differences in patients' quality of life | 1 Month
  First of all, The Cronbach's α coefficient of the EORTC QLQ-C30 patient quality of life questionnaire that is used in this study will be calculated; then the minimum, maximum, median (quartile) and mean (standard deviation) of the quality of life scores of patients of the study group and the control group will be determined; we will use t test to compare the scores to investigate whether two groups are statistically different in each field. Finally, several common influencing factors will be selected to construct a covariance analysis regression model to assess whether the scores of the quality of life of the two groups are statistically different in various fields.
To assess the difference in the quality of life of the subjects (family of patients) 2 months after follow-up management. | 2 Months
  The minimum, maximum, median (quartile) and mean (standard deviation) of the quality of life scores of the family members of the study group and the control group patients after 2 months of follow-up are calculated; T test will be used to compare whether there is a difference in the quality of life score between two groups; then several common influencing factors will be selected to construct a covariance analysis regression model to assess whether the quality of life scores of the two groups of patients are statistically different after 2 months of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital & Institute, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] He Jie, Zhao Ping, Chen Wanqing. China tumor registration report in 2012[M]. Beijing: Military Medical Science Press, 2012:1-302.
- [Background] Borji M, Nourmohammadi H, Otaghi M, Salimi AH, Tarjoman A. Positive Effects of Cognitive Behavioral Therapy on Depression, Anxiety and Stress of Family Caregivers of Patients with Prostate Cancer: A Randomized Clinical Trial. Asian Pac J Cancer Prev. 2017 Dec 28;18(12):3207-3212. doi: 10.22034/APJCP.2017.18.12.3207. PMID 29281868
- [Background] 梁文珍，谭文娟，舒放, 癌症患者家属心理健康状态的调查［J］, 临床 心身疾病杂志，2008，14（2）：136 _ 138
- [Background] 陈冰芳, 实施家属健康教育对鼻咽癌放疗病人生活质量的影响［J］, 护理研究，2010，24，（10c）：2220 _ 2221
- [Background] Greer JA, Jacobs J, Pensak N, MacDonald JJ, Fuh CX, Perez GK, Ward A, Tallen C, Muzikansky A, Traeger L, Penedo FJ, El-Jawahri A, Safren SA, Pirl WF, Temel JS. Randomized Trial of a Tailored Cognitive-Behavioral Therapy Mobile Application for Anxiety in Patients with Incurable Cancer. Oncologist. 2019 Aug;24(8):1111-1120. doi: 10.1634/theoncologist.2018-0536. Epub 2019 Jan 25. PMID 30683710
- [Background] Kim Y, Schulz R. Family caregivers' strains: comparative analysis of cancer caregiving with dementia, diabetes, and frail elderly caregiving. J Aging Health. 2008 Aug;20(5):483-503. doi: 10.1177/0898264308317533. Epub 2008 Apr 17. PMID 18420838
- [Background] Chen W, Sun K, Zheng R, Zeng H, Zhang S, Xia C, Yang Z, Li H, Zou X, He J. Cancer incidence and mortality in China, 2014. Chin J Cancer Res. 2018 Feb;30(1):1-12. doi: 10.21147/j.issn.1000-9604.2018.01.01. PMID 29545714
- [Background] Cohen R, Leis AM, Kuhl D, Charbonneau C, Ritvo P, Ashbury FD. QOLLTI-F: measuring family carer quality of life. Palliat Med. 2006 Dec;20(8):755-67. doi: 10.1177/0269216306072764. PMID 17148530
- [Background] Alnjadat, R. M., Wan Adnan, W. A., & Ismail, Z. (2014). Psychometric properties of the QOLLTI-F questionnaire to assess quality of life in caregivers of cancer patients. Education in Medicine Journal, 6(2).doi:10.5959/eimj.v6i2.217
- [Background] 肖惠敏, 郑建伟, 兰秀燕. 晚期癌症患者生存质量对家庭照顾者生存质量的影响The impact of advanced cancer patients' quality of life on family caregivers' quality of life[J]. 中华护理杂志, 2015, 050(004):415-419
- [Background] 杨理, 刘伟, 邓映, et al. 血液肿瘤患儿家庭照顾者生活质量与家庭环境的相关性分析[J]. 国际护理学杂志, 2018, 37(18):2520-2524
- [Background] Bergman B, Aaronson NK, Ahmedzai S, Kaasa S, Sullivan M. The EORTC QLQ-LC13: a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30) for use in lung cancer clinical trials. EORTC Study Group on Quality of Life. Eur J Cancer. 1994;30A(5):635-42. doi: 10.1016/0959-8049(94)90535-5. PMID 8080679
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Fayers P, Bottomley A; EORTC Quality of Life Group; Quality of Life Unit. Quality of life research within the EORTC-the EORTC QLQ-C30. European Organisation for Research and Treatment of Cancer. Eur J Cancer. 2002 Mar;38 Suppl 4:S125-33. doi: 10.1016/s0959-8049(01)00448-8. PMID 11858978